CLINICAL TRIAL: NCT05736354
Title: Molecular Mechanisms Associated With Breast Implant Complications
Acronym: MMABIC
Status: Recruiting | Type: Observational
Sponsor: Indiana University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Mithun Sinha, Assistant Professor, Indiana University
Other Study IDs: 2003674175; R21AI171932 (NIH); R01AI165958 (NIH)
Record Dates: First submitted 2023-01-17; First posted 2023-02-21 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Breast Implant; Complications; Infection or Inflammation
MeSH Terms: conditions — Infections; Inflammation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Surgically discarded samples (implants, associated capsule, and tissue). For control participants, adipose tissue will be collected which will be removed during implant placement. 20 mL of blood will be collected at the time of pre-operative surgical preparation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- BII Subjects: Subjects with breast implants having BII manifestations.
- Non-BII Subjects: Subjects with breast implants with no reported BII symptoms.
- Subjects without Breast Implants: Subjects without breast implants.

SUMMARY:
Bacterial biofilms cause implant failures, chronic inflammation, and immune polarization. The study investigates the possible role of bacterial biofilm as a factor in the etiology of Breast Implant Illness. Three patient cohorts will be studied (A) Subjects with breast implant with BII manifestations (B) Subjects with breast implants without BII manifestations (C) Subjects without breast implants who underwent breast surgery procedure. Blood, surgically discarded tissue, implants, and associated capsules will be collected through this protocol.

DETAILED DESCRIPTION:
Breast implants were first introduced in 1962. It is estimated that 10 million women worldwide, including three million Americans have breast implants. There has been increased identification of patients experiencing a constellation of symptoms related to their implants. For breast implants, these symptoms are often associated with autoimmune and connective tissue disorders (CTD) and have been referred to as Breast Implant Illness (BII). A growing number of patients 30,000 annually are seeking to have their breast implants removed. In view of the implant associated complications, the US Food and Drug Administration (FDA) has placed a black box warning on breast implants. Limited research has resulted in a void in the prognosis of this surgical problem. Bacterial biofilms are becoming a major concern for medical device implants. Bacterial biofilms cause implant failures, chronic inflammation, and immune polarization. The study investigates the possible role of bacterial biofilm as a factor in the etiology of BII.

This research studies oxilidized lipids (oxylipins). These are metabolities formed as a result of host-biofilm interaction. The presence of oxylipins will be studied in peri-prosthetic tissue post-biofilm infection and in systemic circulation. Oxylipins are immunogenic. Hence, the investigators will also study the abundance of immune cells T cells and macrophages (types and subtypes) and associated cytokines.

ELIGIBILITY:
Inclusion Criteria for breast implant subjects:

* Age greater than or equal to 18 years
* Undergoing removal of breast implant
* Willing and able to comply with protocol instructions

Inclusion Criteria for subjects undergoing breast surgeries (other than implant removal)

* Age greater than or equal to 18 years
* Undergoing breast surgery
* Willing and able to comply with protocol instructions

Exclusion Criteria:

* Individuals who are deemed unable to understand the procedures, risks, and benefits of the study, (i.e., unable to provide informed consent)
* Pregnant females
* Immunodeficiency (HIV/AIDS, SCID)
* Currently on immunosuppressive medications
* Prisoners

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population focuses on females, ages 18 years or older, that are either undergoing removal of breast implants or undergoing breast surgery. Participants must be willing to comply with protocol instructions and possess the mental capabilities to understand the procedures, risks, and benefits of the study. Additionally, participants that are pregnant will not be eligible for participation. Lastly, participants that are deemed immunodeficient or currently taking immunosuppressive medications will be ineligible for participation.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-01-03 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Presence of Biofilm in Breast Tissue | Through study completion, an average of 1 year
  During a clinically scheduled breast surgery, breast tissue specimens will be taken from surgically discarded tissue. The specimens from both breast implant subjects and control subjects (those undergoing breast surgery for a reason other than implant removal) will be analyzed to determine the presence of bacterial biofilm.
Analysis of host-biofilm interaction mediated oxylipins from blood | Through study completion, an average of 1 year
  Prior to a clinically scheduled breast surgery, 20 milliliters of blood will be collected during the pre-operative surgical preparations. The blood samples from both breast implant subjects and control subjects (those undergoing breast surgery for a reason other than implant removal) will be analyzed for host-biofilm interaction mediated oxylipins.
Cytokine analysis will be performed on breast tissue | Through study completion, an average of 1 year
  During a clinically scheduled breast surgery, breast tissue specimens will be taken from surgically discarded tissue. The specimens from both breast implant subjects and control subjects (those undergoing breast surgery for a reason other than implant removal) will undergo cytokine analysis.
Analysis of host-biofilm interaction mediated oxylipins from breast tissue | Through study completion, an average of 1 year
  During a clinically scheduled breast surgery, breast tissue specimens will be taken from surgically discarded tissue. The specimens from both breast implant subjects and control subjects (those undergoing breast surgery for a reason other than implant removal) will undergo oxylipin analysis.

SECONDARY OUTCOMES:
CD4+ Immunological Activation due to Host Implant Interaction | Through study completion, an average of 1 year
  Determining activation of CD4+ immune cells

CONTACTS AND LOCATIONS:
Overall Officials: Mithun Sinha, PhD., Principal Investigator — Indiana University School of Medicine
Locations (3):
- United States (3):
  - IU Health North Hospital, Carmel, Indiana
  - Meridian Plastic Surgeons, Carmel, Indiana
  - IU Health Methodist Hospital, Indianapolis, Indiana